CLINICAL TRIAL: NCT03792698
Title: Preventing Rehospitalization in Lung Transplant Recipients Through mHealth Utilizing Individualized Rehabilitation Prescriptions
Brief Title: Preventing Rehospitalization in Lung Transplant Recipients Utilizing mHealth
Acronym: PERSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Joshua M. Diamond MD,MSCE, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 831322
Record Dates: First submitted 2018-12-14; First posted 2019-01-03 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lung Transplant; Complications
Keywords: Lung Transplantation; Frailty; Readmisson; Physical Therapy; Personalized
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Pre-post intervention study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aidcube utilization (Experimental): Aidcube is a fully customizable, commercially available digital "app"-based platform to deliver home-based pulmonary rehabilitation for patients. On the patient-facing side, patients can view their daily exercise prescription, descriptions and videos demonstrating correct execution of the exercises, document completion of exercises, and message their health-care provider. On the provider-facing side, from over 150 available exercises, surveys, and activities, providers can design a fully-customized exercise prescription. Based on real-time patient feedback, the exercise prescription can be progressed (i.e., advanced and/or modified) by adding repetitions or time to specific exercises or adding new activities. The provider can also message the patient from within the Aidcube environment.
  Interventions: Other: Aidcube digital app-based platform

INTERVENTIONS:
Other: Aidcube digital app-based platform — Use of customizable, patient-specific mHealth home rehabilitation plan

SUMMARY:
Lung transplantation has several important aims: 1) extend survival; 2) relieve disability, and 3) improve health-related quality of life (HRQL) for adults suffering from end-stage lung disease. Advances in medical therapies and changes in the US organ allocation system in 2005 have prioritized lung transplant for sicker and older patients. This achievement has come at substantial cost, including recent trends in recipients towards increased disability, poorer health-related quality of life, and increased longer-term mortality. Additionally, lung transplant recipients have the highest risk of unexpected readmission after the index admission, with published rates of 40-43%. Frailty at the time of discharge is one of the leading factors for readmission. The investigator's belief is that improving access to individualized exercise training plans that are modified based on a patient's progress and needs will greatly improve a transplant recipient's level of physical fitness and independence, and decrease the risk of hospital readmission. This will lead to an overall improvement in a patient's quality of life.

DETAILED DESCRIPTION:
Mission and Specific Aims: Lung transplantation has several important aims: 1) extend survival; 2) relieve disability, and 3) improve health-related quality of life (HRQL) for adults suffering from end-stage lung disease. Advances in medical therapies and changes in the US organ allocation system in 2005 have prioritized lung transplant for sicker and older patients. This achievement has come at substantial cost, including recent trends in recipients towards increased disability, poorer HRQL, and increased longer-term mortality.

Reflecting these trends, lung transplant recipients have the highest risk of unexpected readmission after the index admission among solid organ transplant patients, with published rates of 38-43%. Over the course of the first post-transplant year, the investigators have shown that 60% of lung transplant recipients have a readmission within 30 days of a hospital discharge, of which 30% occur after initial discharge (as above) and 70% occur after a subsequent readmission (2). Each readmission increases the risk for another unplanned rehospitalization as well as long-term mortality, suggesting that this is a particularly vulnerable population.

Over the last year, the investigators performed a single center cohort study to identify risk factors for readmission after index lung transplant discharge. As part of this initiative, the investigators have been evaluating the role of frailty as measured by the Short Physical Performance Battery (SPPB) test. The SPPB is a three-component battery of lower extremity performance, measures that includes gait speed, chair stands, and balance. The investigators have previously demonstrated that frailty is a risk factor for delisting and death among wait listed lung transplant recipients as well as a significant predictor of mortality within the first year after transplant (Figure 1)(3). In a recent single center cohort study of 90 Penn lung transplant recipients, the investigators demonstrated that patients who are frail at index hospitalization discharge based on SPPB are 3.4 times more likely to have an unplanned re-hospitalization within the next 30 days, regardless of whether they are discharged home or to acute rehab. Interestingly, patients are not frail at the time of listing for transplant - frailty develops during the hospital stay for lung transplantation suggesting that physical frailty is dynamic over a short period of time and may be amenable to intervention. The frequent re-admissions, in part due to significant frailty, lead to 1) increased healthcare expenditures (the median professional and hospital payments at Penn for an unplanned hospitalization following discharge was $13048, 2) severely impact the patient's quality of life, and 3) lead to increased mortality.

The investigators have previously found that, among recipients who were frail at discharge and who were enrolled in an intensive outpatient physical therapy program, the median improvement in SPPB was 6 points and 85.7% became not frail (unpublished data). Although this demonstrates that frailty can be reversed in the lung transplant population, the impact of reduced frailty on subsequent readmission has not been evaluated. It remains unknown whether there are other, less resource intensive, mechanisms for improving frailty. The investigator's belief is that improving access to individualize exercise training plans that are modified based on a patient's progress and needs will greatly improve transplant recipient's level of physical fitness and independence, and decrease the risk of hospital readmission. This will lead to an overall improvement in a patient's quality of life. This study, therefore, targets a population of lung transplant recipients at highest risk for readmission and further complications.

Specific Aim: Evaluate the impact of targeted physical therapy rehabilitation plans utilizing a customizable app based interface on the subsequent readmission rates of lung transplant patients at the highest rate of readmission. Patients who are 1) frail at the time of discharge (SPPB≤8) or 2) have already been readmitted after their transplant hospitalization are at the highest risk of subsequent readmission. The investigators hypothesize that targeted, individualized rehabilitation plans will reduce the risk of subsequent readmission.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipient
* SPPB score less than or equal to 9 OR a readmission within 30 days of lung transplant discharge

Exclusion Criteria:

* SPPB >9

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Readmission | one year
  difference in readmission rate over the year prior to the above described intervention with the readmission rate in the setting of Aidcube app utilization

SECONDARY OUTCOMES:
Improved frailty score | one year
  Change in short physical performance battery (SPPB) scores
Health related quality of life | one year
  Change in HRQOL as measured by the Medical Outcomes Survey Short Form 12 (SF12). The SF12 is a 12 question survey designed to assess a subjects mental and physical functioning as well as overall health related quality of life. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Both Physical and Mental Health Composite Scales combine the 12 items in such a way that they compare to a national norm with a mean score of 50.0 and a standard deviation of 10.0. Higher score indicated higher level of functioning.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No